CLINICAL TRIAL: NCT06049706
Title: Priming in Repetitive Transcranial Magnetic Stimulation (TMSr) in the Adjuvant Treatment of Obsessive Compulsive Disorder (OCD)
Brief Title: Priming in Repetitive Transcranial Magnetic Stimulation in the Treatment of Obsessive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suellen Andrade (Other)
Responsible Party: Sponsor-Investigator, Suellen Andrade, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PrimingTMS/OCD
Record Dates: First submitted 2022-07-14; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: priming; supplementary motor area; obsessive-compulsive disorder; transcranial magnetic stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Participants will be divided into 02 groups, each with 16 patients, totaling 32 volunteers: Active - participants who will receive real priming stimulation; Sham - participants who will receive simulated priming stimulation. Participants entered into the study through the eligibility criteria will be randomly allocated in a simple way, at a rate of 1:1.
Who Masked: Participant, Investigator
Masking Description: Duble (Participant, Investigator) All examiners will be blinded to the type of treatment the patient received (active stimulation or sham) and other assessments. Thus, all guidelines established by CONSORT 2010 (Consolidated Standards of Reporting Trials) will be complied with variable control following systematized and countersigned procedures: random sequence generation, allocation concealment, blinding of participants and professionals, blinding of outcome evaluators and attrition bias (loss analysis using the last observation carried forward method)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Priming (TMSr) (Experimental): To apply intervention, it will be used Repetitive Transcranial Magnetic Stimulation Model MagPro R20 (MagVenture Brazil, country Brazil) and the butterfly coil MCF-B70 (MagVenture Brazil, country Brazil).
  Each session will last around 20 minutes, and it will be used a 1 Hz frequency, 1200 pulses/day, with 100% of Motor Threshold, once a day, 5 days a week, for two consecutive weeks.
  Active Priming group participants will be previously stimulated for 10 minutes (20 trains of 5 seconds with intertrain interval of 25 seconds), with 6Hz frequency over Supplementary Motor Area, receiving 80% of Motor Threshold, with a total of 600 stimulations.
  Interventions: Device: Active Priming
- Sham Priming (Sham Comparator): Sham Priming group participants will receive a placebo stimulation for ten minutes, with the same parameters and target area as the active group, they will hear the equipament noise and might feel any sensation in the scalp, but there won't be effective stimulation.
  Interventions: Device: Sham Priming

INTERVENTIONS:
Device: Active Priming — It will be applied an active priming stimulation in the supplementary motor area previously to the main stimulation to analyse if that will enhance the response to TMSr, compared to inactive priming.
  To apply intervention, it will be used Repetitive Transcranial Magnetic Stimulation Model MagPro R20 (MagVenture Brazil, country Brazil) and the butterfly coil MCF-B70 (MagVenture Brazil, country Brazil).
  Each session will last around 20 minutes, and it will be used a 1 Hz frequency, 1200 pulses/day, with 100% of Motor Threshold, once a day, 5 days a week, for two consecutive weeks.
  Active Priming group participants will be previously stimulated for 10 minutes (20 trains of 5 seconds with intertrain interval of 25 seconds), with 6Hz frequency over Supplementary Motor Area, receiving 80% of Motor Threshold, with a total of 600 stimulations.
  Other Names: Priming TMSr
  Arms: Active Priming (TMSr)
Device: Sham Priming — Sham Priming group participants will receive a placebo stimulation for ten minutes, with the same parameters and target area as the active group, they will hear the equipament noise and might feel any sensation in the scalp, but there won't be effective stimulation.
  Arms: Sham Priming

SUMMARY:
Obsessive Compulsive Disorder results in high social impact, affecting quality of life and tending to a chronic course. A considerable proportion of patients, up tp 60%, remain with symptoms even thought treatment is administrated. Therefore, new therapeutic interventions are highly necessary. In this context, repetitive transcranial magnetic stimulation has been used for several psychiatric conditions, including OCD treatment. Moreover, many approaches of neuromodulation seem to reach a better result when used a priming stimulation. In an attemp to optimize particularities of the thecnique applied, this study aims to assess if a priming stimulation with rTMS might impact in a better outcome when compared with rTMS without previous stimulation.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham-controlled clinical trial. Neuropsychological tests and a sociodemographic and clinical questionnaire will be used to assess and characterize the subjects. Participants captured by the Laboratory of Studies in Aging and Neuroscience at the Federal University of Paraíba will be divided into 02 groups, each with 16 patients, totaling 50 volunteers: Active - participants who will receive real priming stimulation; Sham - participants who will receive simulated priming stimulation. Participants entered through the eligibility criteria will be randomly allocated in a simple way, at a rate of 1:1.

In the active priming, the parameters are: frequency of 6 Hz for 10 minutos, 80% do Motor Threshold (MT), 20 trains of 5 seconds, with intertrain interval of 25 seconds, a total f 600 stimulations. The group of innactive priming will have the same parameters, but without active atimulation. After this previous stimulation, all participants will receive the main stimulation: 10 sessions of rTMS, each lasting around 20 minutes, for 5 days a week, during two consecutive weeks.

The target area will be the supplementary motor area. Primary outcome will be assessed by change in Yale-Brown Obsessive Compulsive Scale scores. As secondary outcomes, it will be used HAM-A for anxiety, HAM-D for depression, CGI-S for global clinical impression and SF-36 for quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Being right-handed;
* Age between 18 and 60;
* Diagnose of OCD according to DSM-5;
* Score in YBOCS between 16 and 23;
* No change in dose prescription in the previous 3 months;
* Signature of informed consent term.

Exclusion Criteria:

* Being pregnant;
* Having cognitive deficit;
* Diagnose of drug use disorder;
* In current psychotherapy (or interrupted in less than 3 months);
* Diagnose of severe Major Depression;
* Risk of suicide;
* Patients with metallic implants in the brain;
* Epileptics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive Compulsive Scale | From date of randomization (1 week before intervention beginning) and up to 8 weeks
  It's a 10-item-scale that evaluates the symptoms' severity of Obsessive Compulsive Disorder. Includes five dimensions that evaluate obsessions and compulsions. The ten itens score from 0 (no symptom) to 4 (extreme symptoms), possibly scoring from 0-20 in obsessions' severity, 0-20 in compulsions' severity, with a total 0-40. YBOCS is considered gold standard in evaluating the severity of OCD symptoms.

SECONDARY OUTCOMES:
Change in Hamilton Scale for Depression | From date of randomization (1 week before intervention beginning) and up to 8 weeks
  It's a multidimensional scale which allows evaluating depression symptoms. It will be chosen the variant of 17-item, given that the 21-item doesn't add relevant information for our purposes.
Change in Hamilton Scale for Anxiety | From date of randomization (1 week before intervention beginning) and up to 8 weeks
  A 14-item scale that evaluates both physical and psychological aspects of anxiety
Change in Clinical Global Impression - Scale | From date of randomization (1 week before intervention beginning) and up to 8 weeks
  It's divided into two sub-scales, one that evaluates the severity of disease and one that evaluates clinical improvements. Scores from 1 to 7 (in which 7 refers to worse severity or worse improvement).
Change in Medical Outcomes Study 36 - Item Short Form Health Survey | From date of randomization (1 week before intervention beginning) and up to 8 weeks
  Evaluates quality of life and takes into account 36 items, across 8 dimensions.

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Principal Investigator — Federal University of Paraiba
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No